CLINICAL TRIAL: NCT04853849
Title: Treatment of Overactive Bladder With a Digital Conversational Agent: the MOTIVATION Study
Acronym: MOTIVATION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Renalis (Industry)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CECE2021
Record Dates: First submitted 2021-03-26; First posted 2021-04-21 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Overactive Bladder; Urge Incontinence; Pelvic Floor Disorders
Keywords: Digital therapeutic; Overactive bladder; Urge incontinence; Pelvic floor disorders
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a proof of concept study for a digital therapeutic designed to provide first-line behavioral modification therapy for overactive bladder.

DETAILED DESCRIPTION:
The investigators seek to evaluate a commercial digital therapeutic, called CeCe, designed to provide first-line behavioral modification therapy for overactive bladder (OAB). This digital platform provides daily contact with the user to maximize compliance. It allows a provider to administer behavioral modification treatment while minimizing in-office visits.

The investigators expect that a proportion of participants using Cece will experience significant and satisfactory improvement in their voiding symptoms, to the point where no further treatment is necessary. Others will require additional treatment with the usual therapies such physical therapy and medications, per clinical standards.

Participants will download CeCe to their smart phones and interact with the program for 8 weeks. Participant consent and specific instructions will be provided during study enrollment and through the app. Study outcomes are collected through the program via in-app questionnaires and voiding diaries.

A total of 50 participants will be recruited. They will be compensated a total sum of $175; $50 at completion of an initial set of questionnaires, $50 at completion of 4 week follow-up questionnaires, and $75 at completion of 8 week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of overactive bladder with urgency urinary incontinence, with or without nocturia/nocturnal enuresis
* Symptoms of mixed urinary incontinence if urgency incontinence is the predominant complaint
* Post-void residual <100ml
* English speaking
* Access to a smartphone
* Normal urinalysis without evidence of UTI, gross or microscopic hematuria
* Greater than 6 months since receiving intradetrusor injection of botulinum toxin
* Not currently undergoing sacral neuromodulation therapy
* Not currently receiving pharmacotherapy for overactive bladder

Exclusion Criteria:

* Less than 40 years of age
* Mixed incontinence with predominant stress urinary incontinence symptoms
* Diagnosis of chronic pelvic pain
* symptomatic pelvic organ prolapse
* symptoms of dysuria
* Diagnosis of interstitial cystitis/painful bladder syndrome
* Reported >2 UTI in 6 months or >3 in 12 months
* Do not have access to a smartphone
* Non-English speaking
* Diagnosis of neurogenic bladder
* Gross or microscopic hematuria
* Has diagnosis of dementia, cognitive impairment or other neurologic condition which impairs decision making
* Current Pharmacotherapy or neuromodulation therapy
* Less than 6 months since intradetrusor botulinum toxin injection
* Has decreased mobility or ambulation
* Has post-void residual >100 mL
* Has BMI > 40 kg/m^2
* Inability to voluntarily contract the pelvic floor muscles (a 0/5 in strength).
* Has >4/10 pain with palpation of levator ani, coccygeus, pyriformis, obturator internus or perineal body

Min Age: 40 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Research will be conducted at all University Hospital sites that have a member of the Female Pelvic Medicine and Reconstructive Surgery division seeing patients. This includes UH Richmond, UH Bedford, St. Johns Westshore Medical Center, Landerbook Medical Center, UH Portage Urology, UH Geauga Urology, UHCMC, and UH Westlake. Women 40 years or older with overactive bladder will be screened for and offered study enrollment by the study investigators at each of the above sites.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change of overactive bladder quality of life measure | Baseline, 4 weeks, and 8 weeks
  International Consultation on Incontinence Questionnaire Overactive Bladder Quality of Life questionnaire (ICIQ-OAB-QoL) is a 26 item questionnaire evaluating quality of life (QoL) in patients with overactive bladder. Scores range from 25-160, with greater values indicating increased impact on quality of life.

SECONDARY OUTCOMES:
Change in symptoms of Overactive bladder | Baseline, 4 weeks, and 8 weeks
  OAB-SS is a symptom assessment questionnaire designed to quantify OAB symptoms. The questionnaire consists of 4 questions. The score ranges from 0-15 with higher score indicating more severe OAB symptoms
Change in general health state | Baseline, 4 weeks, and 8 weeks
  SF-36 is a 36 item questionnaire measuring general health. Scores range from 0-100 with higher scores indicating more favorable health state.
Global impression of improvement | At 4 weeks
  The Patient Global Impression of Improvement (PGI-I) is a global index used to rate the response of a condition to a therapy. Scores range from 1-7, with higher values (5-7) indicating higher degree is improvement and lower values (1-3) indicating worse outcomes.
Global impression of improvement | At 8 weeks
  The Patient Global Impression of Improvement (PGI-I) is a global index used to rate the response of a condition to a therapy. Scores range from 1-7, with higher values (5-7) indicating higher degree is improvement and lower values (1-3) indicating worse outcomes.
Change in anxiety | Baseline, 4 weeks, and 8 weeks
  General Anxiety Disorder 7 item (GAD-7) questionnaire is a measure for assessing generalized anxiety disorder. Score ranges from 0-21 with high scores representing more severe depression.
Usability | 8 weeks
  System Usability Scale (SUS) is a 10 item questionnaire for measuring the usability. Scores range from 0-100, with higher scores indicating better usability.
Usability | 8 weeks
  Nelson's Attributes of Usability (NAU) is a 19 item questionnaire measuring usability. Scores range from 0-50, with higher scores indicating better usability
Usability | 8 weeks
  The Chatbot Usability Questionnaire (CUQ) is a 16 item questionnaire measuring usability of a chatbot. Scores range from 0-100, with higher scores indicating better usability
Mobile device proficiency | Baseline
  The Mobile Device Proficiency Questionnaire (MDPQ-16) is a 16 item survey. Scores range from 8.5 - 40, with higher values indicating greater proficiency with mobile devices.

CONTACTS AND LOCATIONS:
Overall Officials: David Sheyn, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown K, Hilton P. The incidence of detrusor instability before and after colposuspension: a study using conventional and ambulatory urodynamic monitoring. BJU Int. 1999 Dec;84(9):961-5. doi: 10.1046/j.1464-410x.1999.00390.x. PMID 10571620
- [Background] Reynolds WS, McPheeters M, Blume J, Surawicz T, Worley K, Wang L, Hartmann K. Comparative Effectiveness of Anticholinergic Therapy for Overactive Bladder in Women: A Systematic Review and Meta-analysis. Obstet Gynecol. 2015 Jun;125(6):1423-1432. doi: 10.1097/AOG.0000000000000851. PMID 26000514
- [Background] Ostaszkiewicz J, Johnston L, Roe B. Timed voiding for the management of urinary incontinence in adults. Cochrane Database Syst Rev. 2004;2004(1):CD002802. doi: 10.1002/14651858.CD002802.pub2. PMID 14973993
- [Background] Ostaszkiewicz J, Johnston L, Roe B. Habit retraining for the management of urinary incontinence in adults. Cochrane Database Syst Rev. 2004;2004(2):CD002801. doi: 10.1002/14651858.CD002801.pub2. PMID 15106179
- [Background] Roe B, Ostaszkiewicz J, Milne J, Wallace S. Systematic reviews of bladder training and voiding programmes in adults: a synopsis of findings from data analysis and outcomes using metastudy techniques. J Adv Nurs. 2007 Jan;57(1):15-31. doi: 10.1111/j.1365-2648.2006.04097.x. PMID 17184371
- [Background] Kandadai P, O'Dell K, Saini J. Correct performance of pelvic muscle exercises in women reporting prior knowledge. Female Pelvic Med Reconstr Surg. 2015 May-Jun;21(3):135-40. doi: 10.1097/SPV.0000000000000145. PMID 25349943
- [Background] Meister MR, Sutcliffe S, Ghetti C, Chu CM, Spitznagle T, Warren DK, Lowder JL. Development of a standardized, reproducible screening examination for assessment of pelvic floor myofascial pain. Am J Obstet Gynecol. 2019 Mar;220(3):255.e1-255.e9. doi: 10.1016/j.ajog.2018.11.1106. Epub 2018 Dec 7. PMID 30527941
- [Background] Stewart WF, Corey R, Herzog AR, et al. Prevalence of overactive bladder in women: results from the NOBLE program. International Urogynecology Journal 2001; 12: pp. S66
- [Derived] Sheyn D, Chakraborty N, Chen YB, Mahajan ST, Hijaz A. Use of a Digital Conversational Agent for the Management of Overactive Bladder. Urogynecology (Phila). 2024 Jun 1;30(6):536-544. doi: 10.1097/SPV.0000000000001428. Epub 2023 Nov 6. PMID 37930265